CLINICAL TRIAL: NCT07135830
Title: Ashwagandha (Withania Somnifera) and Its Effects on Recovery Perceived and Muscle Strength in Male Handball Players: a Randomized Controlled Trial
Brief Title: Ashwagandha (Withania Somnifera) and Its Effects on Recovery Perceived and Muscle Strength in Male Handball Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: JFF
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Strength Training Adaptations; Recovery
Keywords: ashwagandha; strength; recovery; handball

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwaggandha supplementation (Experimental): Participants in this group took one capsule per day containing 600 mg of ashwagandha
  Interventions: Other: Handball training
- Placebo (Placebo Comparator): The placebo group consumed one capsule per day, identical in color and size to the ashwagandha capsules
  Interventions: Other: Handball training

INTERVENTIONS:
Other: Handball training — Athletes will perfrom their regular handball training

SUMMARY:
This study aims to assess the potential recovery and strength effects of male handball players.

ELIGIBILITY:
Inclusion Criteria:

* Handball players competing nationally

Exclusion Criteria:

* Injured athletes
* Female athletes

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Rating of fatigue | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline. Participants' levels of fatigue were measured using the Rating of Fatigue Scale, which includes 10 descriptors ranging from "not fatigue
Perceived soreness | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline. Perceived muscle soreness was evaluated using a 7-point Likert scale, where 0 indicated no soreness and 6 represented severe pain that s
Knee Extension | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline.
Knee Flexion | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline.
Handgrip | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline.

SECONDARY OUTCOMES:
Total Quality Recovery | Evaluations were conducted at three distinct time points: at baseline and at the 4th and 8th days after the baseline.Perceived recovery was evaluated using the Total Quality Recovery (TQR) scale, which ranges from 6 to 20, with endpoints reflecting "very

IPD SHARING:
Plan to Share IPD: Undecided